CLINICAL TRIAL: NCT02263573
Title: Effect of a New Training Protocol: the PEP'C With Constant Load and Intermittent Recovery (PEP'C-R), on Endurance Parameters and Maximal Cardio-respiratory Function Among Sedentary Older Seniors Over 70.
Brief Title: Effect of PEP'C-R on Endurance Parameters and Maximal Cardio-respiratory Function Among Sedentary Older Seniors Over 70
Acronym: PEP'C-R
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: * Interim analysis on 60 randomized subjects showed significant result for the main outcome (VT1)
  * Enrollment difficulty
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5830
Record Dates: First submitted 2014-10-01; First posted 2014-10-13 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Sedentary Lifestyle in Patients Over 70
Keywords: PEP'C-R; Endurance parameters; Maximal cardio-respiratory function; Older seniors; Over 70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEP'C-R (Experimental): Subjects will benefit from one preliminary session and 18 sessions of PEP'C-R, (2 sessions per week for 9.5 weeks).
  Interventions: Other: PEP'C-R
- Control group (Active Comparator): Subjects do not participate in the program PEP'C-R and continue their usual activities at home for 9.5 weeks.
  Interventions: Other: Control group usual activities

INTERVENTIONS:
Other: PEP'C-R — Preliminary session of calibration and tolerance: Test of Borg: determination of VT1 for 10 minutes, 3 min pedaling at 25 W and then 20 minutes pedaling on VT1 determined during the exercise test (ET) -10%.
  Session 1: 30 min of pedaling at constant load VT1 determined during exercise testing (EE) - 10%.
  Session 2 Session 17: increase in the burden of BASE (5 BASE * 5 min: 25 min) by 10% and decrease in relation to the load of the PIC (5 PIC * 1 min: 5 min) to get a cumulative charge of the same session. Changes in heart rate (HR) determine the evolution of sustained loads: a decrease of 10 bpm in heart rate leads to an increase by 10% in the intensity of the base (PIC load remains constant).
  Session 18 = Session 1.
  Arms: PEP'C-R
Other: Control group usual activities — Participants in the control group will not follow the intervention PEP'C-R. They will continue their usual activities for 9.5 weeks and will be assessed before and after this period. After the study, they will be offered the benefit of the conventional program of the PEP'C.
  Arms: Control group

SUMMARY:
The primary purpose of the protocol is to determine the effects of a new program of PEP'C "PEP'C with constant load and intermittent recovery" (PEP'C-R) on endurance parameters of older seniors.

The study hypothesis: the investigators propose that PEP'C-R training offers a significant improvement in endurance parameters for older seniors.

The secondary objectives are to determine the effects of PEP'C-R on maximal cardio-respiratory function, FMD (Flow-mediated dilation), PWV (pulse wave velocity), systolic and diastolic heart function, body composition (measured by impedance), biological, functional and cognitive functioning and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Low physical activity determined using the questionnaire IPAQ in METs (<3).
* Informed about the results of examinations performed at screening visit.
* Subject able to understand the purpose, procedures and risks of the study and give written informed consent.

Exclusion Criteria:

* Contraindications to perform the cardiac stress test and PEP'C-R (Musculoskeletal limitations, Unstabilized heart Failure with chest pain on exertion under maximal medical therapy, ventricular and supraventricular disorders, Acute coronary syndrome within <1 month, Unstabilized respiratory failure or oxygen-dependent)
* Abnormality shown at the cardiac stress test : clinical abnormality (chest pain), electric abnormality (found on ECG), abnormal blood pressure, abnormality of the ventilatory system (bronchospasm, hypoxemia,...)
* Cognitive impairment which exclude PEP'C-R training.
* Current Cancer chemotherapy.
* Visual Impairment which exclude PEP'C-R training.
* Presence of fibromyalgia.
* Subject treated with beta-blockers and other negative chronotropic molecules.
* Acute infection at the time of inclusion.
* Dependent patient.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Change in intensity in W of the first ventilatory threshold (VT1) | From baseline to 9.5 weeks
  Determine the intensity in W of the first ventilatory threshold (VT1) for the experimental group and for the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas VOGEL, MD, PhD, Principal Investigator — CHRU Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

REFERENCES:
- [Derived] Bouaziz W, Schmitt E, Vogel T, Lefebvre F, Lepretre PM, Kaltenbach G, Geny B, Lang PO. Effects of a short-term Interval Aerobic Training Programme with active Recovery bouts (IATP-R) on cognitive and mental health, functional performance and quality of life: A randomised controlled trial in sedentary seniors. Int J Clin Pract. 2019 Jan;73(1):e13219. doi: 10.1111/ijcp.13219. Epub 2018 Jul 2. PMID 29963733